CLINICAL TRIAL: NCT02000349
Title: Comparison of Frozen-thawed Embryo Transfers and Fresh Embryo Transfers With Whole Chromosome Analysis Using Next Generation Sequencing
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Reprogenetics (Industry)
Collaborators: Reproductive Medicine Lab, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Reprogenetics-3.117
Record Dates: First submitted 2013-09-19; First posted 2013-12-04 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Infertility
Keywords: infertility; next generation sequencing
MeSH Terms: conditions — Infertility | interventions — Prostaglandins D; High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Frozen Embryo Transfer with PGD (Experimental): All embryos will be hatched on day 3. Patients will have hatching blastocysts (*) biopsied on day 5 or day 6, embryos will then be vitrified, analyzed by NGS, and will have one or two euploid embryo(s) thawed and transferred on a FET cycle, before noon. If more than two euploid blastocysts are available the one(s) to be transferred will be selected based on morphology (*).
  Interventions: Other: PGD
- Fresh Embryo Transfer with PGD (Experimental): All embryos will be hatched on day 3. Patients will have hatching blastocysts (*) biopsied on day 5, analyzed by NGS, and will have one or two euploid embryo transferred on day 6, in the am. If more than two euploid blastocysts are available the one(s) to be transferred will be selected based on morphology (*). Any morulas developing to hatching blastocyst on day-6 will be also analyzed but vitrified for use in a future cycle.
  Interventions: Other: PGD

INTERVENTIONS:
Other: PGD — PGD using Next generation sequencing
  Other Names: PGD (Preimplantation Genetic Diagnosis); NGS (Next Generation Sequencing)

SUMMARY:
The investigators propose to perform a clinical randomized trial to evaluate the effect of a frozen-thawed embryo transfer and a fresh embryo transfer on pregnancy and implantation rates; with the added benefit of a blastocyst biopsy and whole chromosome analysis by Next Generation Sequencing (NGS).

DETAILED DESCRIPTION:
1. Fresh group: All embryos will be hatched on day 3. Patients will have hatching blastocysts (*) biopsied on day 5, analyzed by NGS, and will have one or two euploid embryo transferred on day 6, in the am. If more than two euploid blastocysts are available the one(s) to be transferred will be selected based on morphology (*). Any morulas developing to hatching blastocyst on day-6 will be also analyzed but vitrified for use in a future cycle.
2. Frozen group: All embryos will be hatched on day 3. Patients will have hatching blastocysts (*) biopsied on day 5 or day 6, embryos will then be vitrified, analyzed by NGS, and will have one or two euploid embryo(s) thawed and transferred on a FET cycle, before noon. If more than two euploid blastocysts are available the one(s) to be transferred will be selected based on morphology (*).

(*) Hatching blastocysts as described by Gardner and Schoolcraft (1999):

ELIGIBILITY:
Inclusion Criteria (pre-stimulation):

* Age up to 42 years

Exclusion Criteria (pre-stimulation):

* MESA and TESE patients
* At least one partner carrier of a chromosomal abnormality
* Egg donor cycle (sperm donor is acceptable)
* Gender selection cycles
* Thaw cycles
* Any patient who cannot have a fresh embryo transfer
* FSH above 12 or AMH less than 1

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 186 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | 8 weeks after replacement
  determining whether a frozen or a fresh embryo transfer will improve implantation rate.

SECONDARY OUTCOMES:
Correlation of Mitochondrial DNA and implantation | When a fetal heartbeat is detected (8 weeks after implantation)
  The second aim of this study is to determine retrospectively if mt DNA content is linked to implantation potential and if that is measurable by NGS. NGS provides the additional advantage that it can measure mitochondrial DNA, which it's content, seems to be inversely correlated with implantation (Fragouli et al 2013, ASRM).

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Munne, PhD, Study Director — Reprogenetics
Locations (1):
- Reproductive Medicine Lab, LLC, Portland, Oregon, United States

REFERENCES:
- [Background] Ata B, Kaplan B, Danzer H, Glassner M, Opsahl M, Tan SL, Munne S. Array CGH analysis shows that aneuploidy is not related to the number of embryos generated. Reprod Biomed Online. 2012 Jun;24(6):614-20. doi: 10.1016/j.rbmo.2012.02.009. Epub 2012 Feb 25. PMID 22503277
- [Background] Cohen J, DeVane GW, Elsner CW, Kort HI, Massey JB, Norbury SE. Cryopreserved zygotes and embryos and endocrinologic factors in the replacement cycle. Fertil Steril. 1988 Jul;50(1):61-7. doi: 10.1016/s0015-0282(16)60009-2. PMID 3384119
- [Background] Cohen J, Wells D, Munne S. Removal of 2 cells from cleavage stage embryos is likely to reduce the efficacy of chromosomal tests that are used to enhance implantation rates. Fertil Steril. 2007 Mar;87(3):496-503. doi: 10.1016/j.fertnstert.2006.07.1516. Epub 2006 Dec 4. PMID 17141767
- [Background] De Vos A, Staessen C, De Rycke M, Verpoest W, Haentjens P, Devroey P, Liebaers I, Van de Velde H. Impact of cleavage-stage embryo biopsy in view of PGD on human blastocyst implantation: a prospective cohort of single embryo transfers. Hum Reprod. 2009 Dec;24(12):2988-96. doi: 10.1093/humrep/dep251. Epub 2009 Sep 21. PMID 19773223
- [Background] Sagoskin AW, Levy MJ, Tucker MJ, Richter KS, Widra EA. Laser assisted hatching in good prognosis patients undergoing in vitro fertilization-embryo transfer: a randomized controlled trial. Fertil Steril. 2007 Feb;87(2):283-7. doi: 10.1016/j.fertnstert.2006.07.1498. Epub 2006 Nov 13. PMID 17094975
- [Background] Fragouli E, Spath K, Alfarawati S, Wells D (2013) Quantification of mitochondrial DNA predicts the implantation potential of chromosomally normal embryos. Fertil Steril, in press (ASRM abstract)
- [Background] Gardner DK and Schoolcraft WB. In vitro culture of human blastocysts. In: Jansen R, Mortimer D. eds. Towards Reproductive Certainty: Fertility and Genetics Beyond 1999. Carnforth, Parthenon Publishin, 1999, 378-88
- [Background] Gutierrez-Mateo C, Colls P, Sanchez-Garcia J, Escudero T, Prates R, Ketterson K, Wells D, Munne S. Validation of microarray comparative genomic hybridization for comprehensive chromosome analysis of embryos. Fertil Steril. 2011 Mar 1;95(3):953-8. doi: 10.1016/j.fertnstert.2010.09.010. Epub 2010 Oct 25. PMID 20971462
- [Background] Hodes-Wertz B, Grifo J, Ghadir S, Kaplan B, Laskin CA, Glassner M, Munne S. Idiopathic recurrent miscarriage is caused mostly by aneuploid embryos. Fertil Steril. 2012 Sep;98(3):675-80. doi: 10.1016/j.fertnstert.2012.05.025. Epub 2012 Jun 7. PMID 22683012
- [Background] Munne S, Wells D, Cohen J. Technology requirements for preimplantation genetic diagnosis to improve assisted reproduction outcomes. Fertil Steril. 2010 Jul;94(2):408-30. doi: 10.1016/j.fertnstert.2009.02.091. Epub 2009 May 5. PMID 19409550
- [Background] SART (2011): https://www.sartcorsonline.com/rptCSR_PublicMultYear.aspx?ClinicPKID=0
- [Derived] Zaat T, Zagers M, Mol F, Goddijn M, van Wely M, Mastenbroek S. Fresh versus frozen embryo transfers in assisted reproduction. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD011184. doi: 10.1002/14651858.CD011184.pub3. PMID 33539543
- [Derived] Coates A, Kung A, Mounts E, Hesla J, Bankowski B, Barbieri E, Ata B, Cohen J, Munne S. Optimal euploid embryo transfer strategy, fresh versus frozen, after preimplantation genetic screening with next generation sequencing: a randomized controlled trial. Fertil Steril. 2017 Mar;107(3):723-730.e3. doi: 10.1016/j.fertnstert.2016.12.022. Epub 2017 Jan 27. PMID 28139240